CLINICAL TRIAL: NCT05480813
Title: Comparison Between Automated and Manual Component Impaction in Total Hip Arthroplasty: Ergonomic and Efficiency Evaluation
Brief Title: Comparison Between Automated and Manual Component Impaction in Total Hip Arthroplasty
Acronym: KINCISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DEO NV (Industry)
Collaborators: BeScored Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KINCISE
Record Dates: First submitted 2022-07-06; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Total Hip Arthroplasty (THA)
Keywords: KINCISE™; Operational efficiency; Ergonomic impaction; Total Hip Arthroplasty (THA)
MeSH Terms: interventions — Efficiency

STUDY DESIGN:
Intervention Model Description: The one participant of the study is an orthopaedic surgeon. He will execute 48 THA procedures during 4 study days. 24 THA procedures will be executed using the automated KINCISE™ impaction system and 24 THA procedures will be executed using a traditional handheld mallet. He will undergo physical and cognitive tests before the OR day, during lunch breaks and after the OR day. Next to that, operational efficiency and ergonomic impaction will be analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prof. Dr. K. Corten (Other): The one participant of the study is an orthopaedic surgeon. He will execute 48 THA procedures during 4 study days. 24 THA procedures will be executed using the automated KINCISE™ impaction system and 24 THA procedures will be executed using a standard mallet. He will undergo physical and cognitive test before and after the OR day and during lunch breaks. Next to that, operational efficiency and ergonomic impaction will be analysed
  Interventions: Device: Automated KINCISE™ impaction system versus handheld traditional mallet; Other: Efficiency and ergonomics analysis and physical assessments

INTERVENTIONS:
Device: Automated KINCISE™ impaction system versus handheld traditional mallet — The KINCISE™ Surgical Automated System (KINCISE) (DePuy Synthes Products, Inc, Warsaw, IN) was developed to replace the handheld mallet traditionally used in total hip arthroplasty (THA). The device is an FDA-approved medical instrument.
Other: Efficiency and ergonomics analysis and physical assessments — Operational efficiency, ergonomic impaction, cognitive/physical/stress level evaluations,

SUMMARY:
This study will investigate and evaluate the ergonomic impaction and the operational efficiency of the KINCISE™ impaction system in comparison with the manual impaction of a handheld traditional mallet in total hip arthroplasty (THA) procedures.

DETAILED DESCRIPTION:
The automated impaction technology of Depuy Sythes (J&J, Warschau), i.e. KINCISE™, can help surgeons impacting the femur in THA surgeries with constant and consistent energy. Furthermore, the bone preparation, implant positioning and implant assembly automate. Next to that, the KINCISE™ is developed to eliminate mallet impaction methods and thus can reduce the physical fatigue of the surgeon during THA procedures, leading to more reproducible and accurate femur manipulation even during the last procedure of the OR day. Two main research questions will be investigated: "Does the KINCISE™ automated impaction lead to a significant reduction in mental and physical fatigue in comparison with mallet impaction?" and "Does the KINCISE™ automated impaction lead to a reduction in OR time?".

Measurements will be executed during 4 OR days. During each OR day exclusively Kincise impaction (N=2) or handheld traditional mallet impaction (N=2) will be performed. The impaction technique will be randomised and the OR setup will be equal in both situations. The one participant in the study is an orthopaedic hip surgeon. He will execute all the THA procedures and undergo all the physical and cognitive tests. The entire study will be assessed by 2 parties of experienced assessors who are not involved in the surgical procedures: BeScored Institute and DEO.

Each OR day, 2 evaluation sessions and 1 mid break session will be held, led by BeScored Institute: in the morning from 06:50am till 08am, during the afternoon from 03:30pm till 04:40pm and during lunch breaks from 11:30am till 12:05pm. Before each morning evaluation session a cognitive task test of 5 minutes will be executed to get familiar with the cognitive tasks of the evaluation sessions. During each evaluation session the following tests will be executed in the same order: psychometric assessments (7 minutes, consisting of 'mindfulness inventory for sport' questionnaire, perfection for stress scale and observed physical fatigue), energy evaluation and stress levels (5 minutes, consisting of heart beat variability measurements, saliva cortisol levels and saliva alfa-amylase levels), cognitive tasks (30 minutes, consisting of Simon test, pattern-comparison test and psychomotor test) and physical tests (20 minutes, consisting of handgrip test, shoulder endurance, planking and isometric mid-thigh pull performance). During the mid break session only the psychometric assessments and cognitive tasks will be executed.

During the THA procedures itself, DEO will evaluate other ergonomics and operational efficiency using the validated DEO Data Collection Platform including datapoints specific to the use of automated and manual impaction, and RULA and REBA methods.

ELIGIBILITY:
Inclusion Criteria:

* Hip surgeon

Exclusion Criteria:

* /

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Cognitive fatigue - Mindfulness Inventory for Sport | 720 minutes
  The surgeon's ability to remain mindful during the working day will be assessed via the Mindfulness Inventory for Sport, adapted for the purpose of this study. Specifically, this questionnaire involves 15 items and 3 dimensions of mindfulness: awareness, non-judgmentally, refocusing. In addition, a modified version of the Perception for Stress Scale will be used before and after. Perceived physical fatigue has also been assessed at rest using a 10-cm visual analogic scale ranging from "Not fatigued at all" to "Very fatigued". Finally, after each physical testing, the participant will be asked to provide a verbal rating of perceived exertion (RPE) using a visual Borg (6-20) scale[26]. RPE was defined as the "perceived difficulty to exert the physical effort before exhaustion".
Cognitive fatigue - Simon Task | 720 minutes
  The Simon task is a selective inhibition task in which the participant is required to respond as quickly and accurately as possible to the color of a stimulus displayed on a screen regardless its spatial location. Then, depending on its left or right location, the user may be required to withdraw an automatic impulse to be able to answer according to the color of the stimulus. The participant will be asked to respond by pressing the appropriate left or right buttons according to the color of a circle delivered either to the left or to the right of the white gaze-fixation cross. The task includes two equiprobable trial types: the congruent trials during which the spatial location of the stimulus corresponded to the task-relevant aspect of the stimulus, and the incongruent trials in which the spatial location of the stimulus corresponded to the opposite spatial location of the response.
Cognitive fatigue - Pattern-comparison task | 720 minutes
  A pattern-comparison task will also be carried out to assess the surgeon's ability to visually identify anomalies, equipment failures, compliance checks, etc. throughout a surgery. Specifically, in order to test the surgeon's ability to quickly determine the compatibility (similarity) and incompatibility (dissimilarity) of stimuli, a visual comparison task will be performed. The aim will be to respond via the computer keyboard to the convergent dimension of 2 images displayed on the screen for 30 trials, and then to the non-convergent dimension for another 30 trials, in a time lapse of 1.5 sec per trial.
Cognitive fatigue - Psychomotor task | 720 minutes
  The effectiveness of the and surgeon's motor control will be assessed to consider whether careful manual interventions could potentially be affected by both surgical conditions (Kincise automated impaction vs handheld impaction). A psychomotor task will therefore be formed with the instruction to follow, via a computer mouse, the predictable movement of a light spot on the screen. One minute of evaluation will be carried out, with the time of contact with the light target and the average distance to this target as variables of interest.
Physical fatigue - | 720 minutes
  A plank to fatigue test (PFT) will be used to assess lumbar muscle fatigue. Between experimental sessions, the same distance between the 2 feet, between the 2 elbows and between the hip and the floor, will be required for each participant. The distance between the hip and the floor shall serve as the measure of exhaustion. Exhaustion is declared when the distance between the participant's hip and the floor is reduced by more than 2 cm for more than 5 sec.
Physical fatigue - Shoulder endurance | 720 minutes
  Shoulder endurance and deltoideus anterior muscle fatigue will be assessed via light weightlifting. In particular, the participant will be required to maintain a 3 kg weight in front of him, with the arms stretched out (perpendicular to the trunk, 90° adduction) and during 3 periods of 10 sec interspaced with 10-sec resting periods.
Physical fatigue - Handgrip test | 720 minutes
  A handgrip test will be carried out using a hand dynamometer (microFET® Digital HandGRIP Dynamometer, USA). This shall enable us to assess the strength decline of the flexor's muscles of the participant's dominant hand. Ten repeated maximal voluntary contractions shall be performed in 20 sec (i.e., 1 contraction every 2 sec).
Physical fatigue - Isometric mid-thigh pull test | 720 minutes
  an Isometric Mid-Thigh Pull Performance (IMTPP) will be used as a measure of thighs strength of endurance. The posture of this exercise is characterized by the two right angles formed by the body, one at the hips and one at the knees. The participant will also be required to keep their arms stretched out in front of them until exhaustion to avoid compensation movements.
Stress - Salivary cortisol & alpha-amylase | 720 minutes
  We will observe the variations of both salivary cortisol and alpha-amylase in this study at different timepoints. On the morning of each experimental day and at the end of the surgery, the surgeon will provide a 4-mL saliva sample via passive drool. The samples will be obtained in a fasted-state at 5:00 AM and at 4:40 PM and will be promptly frozen at -80°C
Operational efficiency | 28 hours
  Efficiency will be assessed using OR time, by comparing the OR days and procedures where the KINCISE tool or the mallet is used.
  A granular analysis from the timestamps will be conducted using standard descriptive statistics. Additionally, the impaction process will be further analyzed, broken down into parts.
Ergonomic impaction | 28 hours
  Measurement of weight of Kincise and mallet, audio of impaction (Kincise vs mallet) and the surgeon's posture assessment using RULA and REBA method will be combined to report ergonomic impaction on the surgeon by DEO

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Dille, Study Director — DEO NV
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No